CLINICAL TRIAL: NCT06081959
Title: A Randomized, Open-label, Multicenter Phase 3 Study of SKB264 Versus Treatment of Physician's Choice (TPC) in Patients With Unresectable Locally Advanced, Recurrent or Metastatic HR+/HER2- Breast Cancer Who Had Failed at Least One Line of Chemotherapy
Brief Title: Study of SKB264 for Locally Advanced, Recurrent or Metastatic HR+/HER2- Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-Ⅲ-10
Record Dates: First submitted 2023-10-07; First posted 2023-10-13 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin; Capecitabine; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SKB264 for injection (Experimental)
  Interventions: Drug: SKB264
- Treatment of Physician's Choice (Active Comparator): Eribulin, capecitabine, gemcitabine or vinorelbine will be administered and managed according to the investigator's clinical judgment, guided by clinical practice.
  Interventions: Drug: Eribulin; Drug: Capecitabine; Drug: Gemcitabine; Drug: Vinorelbine

INTERVENTIONS:
Drug: SKB264 — IV infusion on day 1 and Day 15 of each 28 day cycle
  Arms: SKB264 for injection
Drug: Eribulin — 1.4 mg/m2, IV infusion on day 1 and Day 8 of each 21 day cycle
  Arms: Treatment of Physician's Choice
Drug: Capecitabine — 1000-1250 mg/m2, po, bid, from day 1 to Day 15 of each 21 day cycle
  Arms: Treatment of Physician's Choice
Drug: Gemcitabine — 1000 mg/m2, IV infusion on day 1 and Day 8 of each 21day cycle
  Arms: Treatment of Physician's Choice
Drug: Vinorelbine — 25 mg/m2, IV infusion on day 1 and Day 8 of each 21 day cycle
  Arms: Treatment of Physician's Choice

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SKB264 in patients with unresectable locally advanced, recurrent, or metastatic HR+/HER2- breast cancer.

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter Phase 3 clinical study to evaluate SKB264 monotherapy versus Treatment of Physician's Choice (TPC) in subjects with unresectable locally advanced, recurrent, or metastatic HR+/HER2- breast cancer who had failed at least one line of systemic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥ 18 to ≤ 75 years at the time of signing the ICF;
* Histologically and/or cytologically confirmed HR+/HER2- breast cancer based on pathology reports on recent biopsy specimens or other pathological samples;
* Patients who had failed at least one line of systemic chemotherapy in unresectable locally advanced, recurrent, or metastatic stage;
* Patients with at least one measurable lesion per RECIST 1.1 criteria; those with only skin or bone lesions cannot be included;
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1;
* Expected survival ≥ 12 weeks;
* Adequate organ and bone marrow function;
* Patients who are eligible for a chemotherapy regimen in the control group;
* Female patients of childbearing potential and male patients with partners of childbearing potential who use effective medical contraception from the time of signing the informed consent form until 6 months after the last dose;
* Patients who voluntarily participate in the study and sign the ICF, and able to comply with the visit and related procedures stipulated in the plan.

Exclusion Criteria:

* Patients with a history of central nervous system (CNS) metastases or current CNS metastases；
* Patients with other malignancies (except cured basal or squamous cell skin cancer or carcinoma in situ of the cervix) within 3 years prior to the first dose;
* Patients with any cardio cerebral Vascular disease or cardio cerebral vascular risk factors may affect investigational treatment;
* Uncontrollable systemic diseases assessed by the investigator;
* History of (noninfectious) interstitial lung disease (ILD)/noninfectious neumonitis requiring steroid therapy and current ILD/noninfectious pneumonitis, or ILD/noninfectious pneumonitis at screening that cannot be excluded by imaging;
* Clinically serious lung injuries caused by lung diseases;
* Patients with active chronic Inflammatory bowel disease, gastrointestinal obstruction, severe ulcer, gastrointestinal perforation, abdominal abscess or acute gastrointestinal bleeding;
* Toxicities from prior anti-tumor therapy not recovering to ≤ Grade 1;
* Active hepatitis B or hepatitis C;
* Human immunodeficiency virus (HIV) antibody test positive or a history of acquired immunodeficiency syndrome (AIDS), known active syphilis infection;
* Known allergy or hypersensitivity to SKB264, or the excipients of SKB264;
* Prior TROP2 targeted therapy, prior topoisomerase I inhibitor therapy, including antibody-drugconjugate(ADC) therapy;
* Patients who received major surgeries 4 weeks prior to the first dose of study treatment or planned to receive major surgeries during the study ;
* Patients with concomitant infections requiring systemic antibiotic therapy within 2 week prior to the first dose of study treatment;
* Patients who have received live vaccines within 30 days prior to the first dose, or are scheduled to receive live vaccines during the study;
* Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) assessed by BIRC per RECIST 1.1. | up to 24 months
  PFS, defined as the time from randomization to PD or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | up to 24 months
  OS, defined as the time from randomization to death
Progression-free survival (PFS) assessed by the investigators per RECIST V 1.1 | up to 24 months
  PFS, defined as the time from randomization to PD or death, whichever occurs first.
Objective Response Rate (ORR) | up to 24 months
  The percentage of patients with CR and PR assessed by BIRC and investigators per RECIST v 1.1
Disease Control Rate (DCR) | up to 24 months
  The percentage of patients who have achieved CR，PR and SD assessed by BIRC and investigators per RECIST v 1.1
Duration of Response (DoR) | up to 24 months
  From the date that response criteria are first met to the first occurrence of PD as determined by BIRC and investigators per RECIST v1.1 or death from any cause, whichever occurs first
Quality of life of patients evaluated using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) scale | Up to 2 years
  To assess the impact of SKB264 on disease related symptoms and health related quality of life (HRQoL) in this patient population
AEs and SAEs | AEs should be observed and recorded from signing the ICF until 30 days after the last dose. AEs occurring 30 days after the last dose are not required to be actively collected by the investigator.
  Incidence and severity of AEs and SAEs (per CTCAE 5.0), and clinically significant abnormal laboratory findings

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality, China